CLINICAL TRIAL: NCT02394457
Title: Cosyntropin Versus Epidural Blood Patch (EBP) for Treatment of Treatment of Post Dural Puncture Headache (PDPH)
Brief Title: Cosyntropin Versus Epidural Blood Patch (EBP) for Treatment of Treatment of Post Dural Puncture Headache
Acronym: PDPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NMCSD.2006.0026
Record Dates: First submitted 2015-02-18; First posted 2015-03-20 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Postdural Puncture Headache
Keywords: Postdural puncture headache; Epidural Blood Patch; Cosyntropin; PDPH; Regional anesthesia; Lumbar puncture; ACTH; Tetracosactin
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Cosyntropin; Blood Patch, Epidural

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Cosyntropin Group A (Experimental): Cosyntropin 500 mcg in 1000cc Normal Saline
  Interventions: Drug: Cosyntropin
- Epidural Blood Patch Group B (Active Comparator): Epidural Blood Patch and I000cc Normal Saline
  Interventions: Procedure: Epidural Blood Patch

INTERVENTIONS:
Drug: Cosyntropin — Intravenous Drug Infusion over 1 hour and a half
  Other Names: Tetracosactin
  Arms: Intravenous Cosyntropin Group A
Procedure: Epidural Blood Patch — Blood drawn from subject and then same Blood placed into Epidural space by anesthesia personnel.
  Other Names: Blood patch
  Arms: Epidural Blood Patch Group B

SUMMARY:
PDPH is a common problem after either intentional or unintentional Dural puncture. It is especially common in young female patients and in patients undergoing Lumbar Puncture using the typical kit containing large 20 gauge needles (1).

Hypothesis is that Cosyntropin therapy is at least as effective as current conservative therapy (caffeine/fluid) and/or Epidural Blood Patch.

Patients will be randomly assigned to undergo either: (1) EBP with IVF therapy or (2)Cosyntropin IV with IVF therapy. Endpoints will be a pain score that is given prior to the procedure, Emergency Department (ED) discharge pain score and post procedural day (PPD) day 1, day 3 and day 7 pain and functional levels. Patients in Cosyntropin arm of the study may request crossover to EBP at anytime after a 24 hour assessment period is completed per Standard of Care for treatment of PDPH, in order to ensure no undue distress is placed on the patient in order to complete this study.

Current treatments consist primarily of non-invasive treatment with intravenous fluids and caffeine therapy and invasive treatment by Epidural Blood Patch. Efficacy of Caffeine 300mg IV bis in die (BID) x 1d doses is approximately 70% (2). However this therapy has been linked to post-treatment seizures. EBP was originally thought to be 90% effective with repeat treatment efficacy approaching >96%. However more recent studies by Taivainen et al (3) have shown only a 61% rate of permanent cure. Additionally, EBP are contraindicated in patients with signs of increased intra-cranial pressure (ICP), coagulation issues, signs/symptoms of Central Nervous System (CNS) /systemic infection or local infection at the site of the EBP, thus resulting in decreased utility. Complications are also quite serious ranging from meningitis, spinal hematoma, repeat dural puncture, localized infection and vagal response to the procedure. EBP are not typically performed until after conservative measures have failed which leads to further prolongation of the patients decreased functional status and pain. Additionally, the cost of both treatments is substantial considering prolonged ED visits for conservative treatments often followed by the time and expense of an EBP.

The goal of this investigation is to aid in the confirmation of case reports advocating the economy, efficacy and safety of synthetic Adrenal CorticTropin Hormone (ACTH) as a treatment of PDPH (4,5,6,7,8,9).

DETAILED DESCRIPTION:
PDPH is a common problem after either intentional or unintentional Dural puncture. It is especially common in young female patients and in patients undergoing Lumbar Puncture using the typical kit containing large 20 gauge needles (1).

Current treatments consist primarily of non-invasive treatment with intravenous fluids and caffeine therapy and invasive treatment by Epidural Blood Patch. Efficacy of Caffeine 300mg IV BID x 1d doses is approximately 70% (2). However this therapy has been linked to post-treatment seizures. EBP was originally thought to be 90% effective with repeat treatment efficacy approaching >96%. However more recent studies by Taivainen et al (3) have shown only a 61% rate of permanent cure. Additionally, EBP are contraindicated in patients with signs of increased ICP, coagulation issues, signs/symptoms of CNS/systemic infection or local infection at the site of the EBP, thus resulting in decreased utility. Complications are also quite serious ranging from meningitis, spinal hematoma, repeat dural puncture, localized infection and vagal response to the procedure. EBP are not typically performed until after conservative measures have failed which leads to further prolongation of the patients decreased functional status and pain. Additionally, the cost of both treatments is substantial considering prolonged ED visits for conservative treatments often followed by the time and expense of an EBP.

The goal of this investigation is to aid in the confirmation of case reports advocating the economy, efficacy and safety of synthetic ACTH as a treatment of PDPH (4,5,6,7,8,9).

After patients receive and sign an informed consent form (ICF) Patients will be randomly assigned to undergo either: (1) EBP with IVF therapy or (2)Cosyntropin IV with IVF therapy. Endpoints will be a pain score that is given prior to the procedure, ED discharge pain score and post procedural day (PPD) day 1, day 3 and day 7 pain and functional levels. Patients in Cosyntropin arm of the study may request crossover to EBP at anytime after a 24 hour assessment period is completed per Standard of Care for treatment of PDPH, in order to ensure no undue distress is placed on the patient in order to complete this study.

Investigational New Drug (IND) Exemption for use of Cosyntropin.

Research Objective: To develop an efficacious and cost effective alternative to Epidural Blood Patch and Caffeine therapy for Postdural Puncture Headache.

Two Study Groups: (1) Group A - Cosyntropin 500 mcg in 1000 mili-liters Normal Saline (NS) run over 1 hour (2) Group B - Epidural Blood Patch and 1000 mili-liters NS

* 1liter NS run over 1 hour while waiting for call team to place Epidural Blood Patch
* Std Epidural Kit using 18g tuohy needle to Loss of Resistance (LOR) with providers preferred medium
* Max 20 cc of sterile blood in epidural space with amount dictated by either 20cc or sig pain/pressure
* Pt supine for 30 minutes post procedure

Randomization Procedures: Computer generated random number list with even numbers receiving Cosyntropin and odd numbers receiving traditional epidural blood patch.

Methods and Materials: After referral to an Anesthesiologist and confirmation of PDPH diagnosis, patient will be randomized to either Cosyntropin or Epidural Blood Patch assuring they are negative for pregnancy. If enrolled in Cosyntropin arm a bag of premixed (by pharmacy) Cosyntropin 500mcg in a 1 liter Normal Saline bag of Intravenous Fluid will be run over 1 hour. Please see above for further details. Additionally, there will be a telephone follow-up questionnaire performed by a person not directly involved with the study to collect data as described above.

Standard of Care: Patients are evaluated by the ED, clinic, labor deck or pre-op area and if PDPH is suspected patient is offered and given conservative treatment with intravenous caffeine. If this treatment fails and/or the patient requests it, the Anesthesia team is notified for possible EBP.

Experimental Procedure: Randomly selected patients will receive Cosyntropin 500mcg IV in 1 liter NS vs EBP

Research Material Collected: Verbal Analogue Scale scores and improvement in functional status. Pt's will be identified by a Patient ID number which will not be the same as the patient's hospital Identification (ID) or Social Security Number (SSN). Contact information will be kept on a separate patient tracking sheet (see attached) and kept electronically on a password protected computer.

Subject Recruiting: All patients meeting inclusion requirements will be offered enrollment at time of diagnosis/treatment.

Justification of Subject Population: Patient's with PDPH often have significant pain levels and subsequent decreases in function. Recent literature notes decreased efficacy of invasive Epidural Blood Patches. Alternate, less invasive techniques, could decrease time to relief and allow treatment patients with contra-indications to Epidural Blood Patch.

Risks: Local Infection, meningitis, allergic reaction, spinal hematoma, nerve damage, paralysis, failure of procedure, new dural puncture. Incidence of adverse events will be tracked.

1. Justification of Risks- Control arm is current standard of care for this patient population. Experimental group utilizes a medication that has a very low risk profile. This medication is often used in the ICU setting on the most critical ill without increased risk.
2. Minimization of Risks- Control arm is current standard of care. Experimental group will be treated in monitored settings of either the Emergency Department, Post- Anesthesia Care Unit (PACU) or L&D PACU
3. Medical Monitor- A medical Monitor will be appointed

Benefits: Optimization of pain control for patients with PDPH. Will provide an alternative method to treat those patients with PDPH who have contra-indications to EBP. Will significantly reduce cost/personnel for treatment of PDPH and give options to medical providers in remote regions of care without the training/equipment to perform EBP.

Statistical Analysis: Data analysis will be accomplished using descriptive and inferential statistics. Demographic data will be analyzed using Student's t-test. Frequency data will be compared with the Chi-square test. A student's t-test will be used to compare the verbal pain scores. The satisfaction scores will be compared with a Mann-Whitney U test. A p-value of < 0.05 will be considered significant. All analysis will be performed utilizing Intention-to-Treat analysis and clearly state in the results section the number of persons that switch from the cosyntropin group to epidural blood patch therapy. The efficacy of the EBP for the study group and for this "crossover" group will also be noted.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older,
2. Diagnosed by Anesthesia provider as having PDPH
3. Agrees to participation in study

Exclusion Criteria:

1. In-patient status and/or unstable medical condition
2. Patient's contraindication to EBP: Local infection at injection site, systemic infection, hemodynamically unstable, severely hypovolemic
3. Patient's contraindication to EBP: Known or past reaction to natural ACTH or Cosyntropin
4. Signs or symptoms of ICP such as Mental Status changes, Bradycardia and hypertension
5. Congestive Heart Failure
6. Patient refusal to participate
7. Current Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hanling, MD, Principal Investigator — NavalMCSD Pain Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] VANDAM LD, DRIPPS RD. Long-term follow-up of patients who received 10,098 spinal anesthetics; syndrome of decreased intracranial pressure (headache and ocular and auditory difficulties). J Am Med Assoc. 1956 Jun 16;161(7):586-91. doi: 10.1001/jama.1956.02970070018005. No abstract available. PMID 13318967
- [Background] Sechzer PH, Abel L. Post-spinal anesthesia headache treated with caffeine. Evaluation with demand method. Part I. Curr Therap Res 1978; 24:307-12.
- [Background] Taivainen T, Pitkanen M, Tuominen M, Rosenberg PH. Efficacy of epidural blood patch for postdural puncture headache. Acta Anaesthesiol Scand. 1993 Oct;37(7):702-5. doi: 10.1111/j.1399-6576.1993.tb03793.x. PMID 8249562
- [Background] Collier BB. Treatment for post dural puncture headache. Br J Anaesth. 1994 Mar;72(3):366-7. doi: 10.1093/bja/72.3.366-c. No abstract available. PMID 8130064
- [Background] Foster P. ACTH treatment for post-lumbar puncture headache. Br J Anaesth. 1994 Sep;73(3):429. doi: 10.1093/bja/73.3.429-a. No abstract available. PMID 7946882
- [Background] Carter BL, Pasupuleti R. Use of intravenous cosyntropin in the treatment of postdural puncture headache. Anesthesiology. 2000 Jan;92(1):272-4. doi: 10.1097/00000542-200001000-00043. No abstract available. PMID 10638928
- [Background] Gupta S, Agrawal A. Postdural puncture headache and ACTH. J Clin Anesth. 1997 May;9(3):258. doi: 10.1016/s0952-8180(97)00042-1. No abstract available. PMID 9172038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 were consented, of these 28 patients met study criteria and were randomized
Period: Overall Study
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Started | 15 | 13
Completed | 15 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Full Range); unit: years] | 29.2 [18 to 65] | 26.9 [18 to 65] | 28.05 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 5 | 11
Pain [Number; unit: units on a scale] — Pain was measured 1-10 scale with 10 representing the highest level of pain, number reported was the mean
  units on a scale | 8.53 | 8.50 | 17.03
Function [Mean (Full Range); unit: units on a scale] — self-reported function scores were 1-10 with 10 representing the greatest impairment to function
  units on a scale | 7.4 [1 to 10] | 7.17 [1 to 10] | 7.29 [1 to 10]
Positional Headache [Number; unit: participants] — measure to obtain headache history was considered positive if the patient reported any previous diagnosis of recurrent headaches or previous post dural headache
  participants | 14 | 11 | 25
Nausea/Vomiting [Number; unit: participants] — measure describes number of patients who reported positive for nausea/vomiting
  participants | 10 | 11 | 21
Neck Stiffness [Number; unit: participants] — measure describes number of patients who reported positive for neck stiffness
  participants | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Headache Pain Score
Description: Numerical 0-10 (0 no pain, 10 worst pain)
Time Frame: 1 day post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Number analyzed (Participants) | 15 | 13
units on a scale | 6.67 (7.56) | 2.33 (2.74)

2. Primary Outcome: Headache Pain Score
Description: Numerical 0-10 (0 no pain, 10 worst pain)
Time Frame: 3 days post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Number analyzed (Participants) | 15 | 13
units on a scale | 3.13 (2.01) | 2.36 (2.47)

3. Primary Outcome: Headache Pain Score
Description: Numerical 0-10 (0 no pain, 10 worst pain)
Time Frame: 7 days post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Number analyzed (Participants) | 15 | 13
units on a scale | 1.93 (1.84) | 1.82 (1.86)

4. Secondary Outcome: Functioning Score
Description: Functional score 0-10 (0 being able to function all tasks of daily living, 10 not able to complete activities of daily living (ADLs)
Time Frame: 1 day post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Number analyzed (Participants) | 15 | 13
units on a scale | 6.53 (1.35) | 2.00 (2.83)

5. Secondary Outcome: Functioning Score
Description: Functional score 0-10 (0 being able to function all tasks of daily living, 10 not able to complete ADLs
Time Frame: 3 day post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Number analyzed (Participants) | 15 | 13
units on a scale | 3.20 (1.81) | 2.09 (2.34)

6. Secondary Outcome: Functioning Score
Description: Functional score 0-10 (0 being able to function all tasks of daily living, 10 not able to complete ADLs
Time Frame: 7 day post procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Number analyzed (Participants) | 15 | 13
units on a scale | 2.14 (1.03) | 1.64 (2.35)

ADVERSE EVENTS:
Arm/Group | Intravenous Cosyntropin Group A | Epidural Blood Patch Group B
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13

LIMITATIONS AND CAVEATS:
Subjects treated with cosyntropin could also receive EBP.Lack of description of patient activity level on follow up.Functional scoring tool not validated.Cost analysis & system utilization not captured.Variations in clinical judgment.Lack of blinding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No